CLINICAL TRIAL: NCT07357233
Title: Impact Of Manual-Less Root Canal Instrumentation Versus Conventional Rotary Instrumentation On Post Operative Pain And Level Of Neuropeptides: Randomized Controlled Clinical Trial
Brief Title: Comparison Between Two Instrumentation Techniques on Postoperative Pain and Level of Neuropeptides
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 928971
Record Dates: First submitted 2025-12-20; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Post Operative Pain
Keywords: manual-less technique; Substance p; CGRP; root canal treatment; irreversible pulpitis; controlled memory; apical fluids; Elisa; Time
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual-less (Experimental): Canals preparation with rotary dota files escaping scouting and glide path step.
  Interventions: Other: Manual-less
- control (Experimental): Canal preparation with rotary dota files with prior scouting and glide path with hand files.
  Interventions: Other: Conventional technique

INTERVENTIONS:
Other: Manual-less — Canals preparation with rotary dota files escaping scouting and glide path step
  Arms: manual-less
Other: Conventional technique — Canal preparation with rotary drill files, with prior scouting and glide path with hand files.
  Arms: control

SUMMARY:
General aim: assessment of post operative pain and time of preparation with the execution of manual-less technique and conventional technique.

Specific aim: correlation between post operative pain and release of Substance P and Calcitonin gene-related peptide.

DETAILED DESCRIPTION:
Background: Post-operative pain (POP) remains a significant challenge after root canal treatment. A recent approach emphasizes objective pain assessment by measuring neuropeptides like substance P (SP) and calcitonin gene-related peptide (CGRP). Rotary nickel-titanium (NiTi) instruments have largely replaced manual stainless-steel files, improving efficiency, maintaining original root canal anatomy and reducing errors. Advances such as controlled memory (CM) files help minimize debris extrusion, potentially lowering POP. A fully rotary approach, eliminating the need for manual scouting and glide path creation, could offer a faster, more predictable alternative. This approach could be named as manual-less technique.

Aim: This study compares between manual-less instrumentation technique (excluding scouting and glide path step) versus conventional rotary instrumentation technique on the post operative pain and release of SP and CGRP.

Materials and methods: A total of 34 permanent molars with symptomatic irreversible pulpitis and apical periodontitis will be included in this study. They will be randomly divided into 2 groups (n=17): group I(manual-less): canal preparation using Dota rotary files escaping scouting and glide path step and Group II (conventional): canal preparation using Dota rotary files with prior scouting and glide path with hand files. Elisa analysis will be done for measuring level of SP and CGRP before and after instrumentation.

Analysis: All data will be collected and statistically analyzed with the appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic irreversible pulpitis and apical periodontitis in mandibular molars with closed apex.(17)
2. Healthy males and females (Category: American Society of Anesthesiologists class I).
3. Age of patients range from 18 to 50 years old.
4. Those who could understand the use of the numeric rating scale (NRS) for pain.
5. In cases where radiographs show no root resorption or abnormal anatomy.
6. Patients with good oral hygiene and free from periodontal diseases.

Exclusion Criteria:

1. Allergy to anesthetics.
2. Pregnancy
3. Unrestorable teeth.
4. Patient on analgesics.
5. Prescence of root resorption or abnormal anatomy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in post operative pain | 6 hours,12 hours,24 hours,48 hours,72 hours
  Numeric rating scale ranges from zero to 10. zero means no pain and 10 means severe pain.

SECONDARY OUTCOMES:
correlation between post operative pain and release of Substance P and Calcitonin gene-related peptide. | first sample in the first visit immediatly post instrumentation ,second sample in the second visit72hr
  ELISA Kit will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt